CLINICAL TRIAL: NCT02746744
Title: RItuximab Versus FUmarate in Newly Diagnosed Multiple Sclerosis. A Randomized Phase 3 Study Comparing Rituximab With Dimethyl Fumarate in Early Relapsing-Remitting Multiple Sclerosis and Clinically Isolated Syndrome.
Brief Title: RItuximab Versus FUmarate in Newly Diagnosed Multiple Sclerosis.
Acronym: RIFUND-MS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Anders Svenningsson (Other)
Responsible Party: Sponsor-Investigator, Anders Svenningsson, MD PhD, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EudraCT 2015-004116-38
Record Dates: First submitted 2016-04-18; First posted 2016-04-21 (Estimated); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Rituximab; Dimethyl Fumarate; Sodium Chloride

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Rituximab (Experimental): Infusion of Mabthera/Rituximab every 6 months
  Interventions: Drug: Rituximab
- Dimethyl Fumarate (Active Comparator): Intake of Tecfidera/Dimethyl Fumarate daily acc. to clinical practice.
  Interventions: Drug: Dimethyl fumarate; Drug: Sodium Chloride solution
- Sodium Chloride solution (Sham Comparator): Sham infusion with sodium chloride solution for the Tecfidera/Dimethyl Fumarate arm every 6 months (so that the examining physician will be blinded)
  Interventions: Drug: Dimethyl fumarate; Drug: Sodium Chloride solution

INTERVENTIONS:
Drug: Rituximab — Infusion of Mabthera/Rituximab every 6 months
  Other Names: Mabthera
  Arms: Rituximab
Drug: Dimethyl fumarate — Intake of Tecfidera/Dimethyl Fumarate daily acc. to clinical practice.
  Other Names: Tecfidera
  Arms: Dimethyl Fumarate; Sodium Chloride solution
Drug: Sodium Chloride solution — Placebo/Sham infusion every 6 months so that the examining physician (blinded) should not know which patient gets Mabthera or Tecfidera
  Other Names: Sodium Chloride
  Arms: Dimethyl Fumarate; Sodium Chloride solution

SUMMARY:
A randomized phase 3 study comparing Rituximab with Dimethyl Fumarate in early Relapsing-Remitting Multiple Sclerosis and Clinically Isolated Syndrome.

DETAILED DESCRIPTION:
This is a prospective randomised phase 3 study comparing a novel treatment protocol of Rituximab with a present first line disease modifying drug regarding both clinical, radiological and biochemical parameters. This will be measured via clinical investigations, MRI and Cerebrospinal fluid analyses. Each patient will have one treating physician responsible for all ongoing medical questions and decisions regarding continuation in the study and one examining physician performing the blinded Expanded Disability Status Scale examination and assessments of exacerbations. The coordinating nurse will administer the study-related tests and administer the rituximab infusions. In order to keep the examining physician blinded the patients receiving disease modifying drug will receive infusions with sodium chloride solution at the same interval as the rituximab arm is receiving. In both instances an opaque cover bag will shield the content of the infusion solution. In this case the examining physician will not be able to identify rituximab patients in case of accidental meetings on the neurology unit.

Randomisation will be performed via a randomisation module in the national Swedish MS registry. The patients will be randomised in a 1:1 ratio and receive their treatments in accordance with clinical practice. Thus, the study will mimic the real-life situation in which the treatments will be administered which involves both positive and negative consequences. As positive consequence the result of the study will have a high degree of validity in relation to expected outcome in clinical practice. As negative consequence there may be psychological effects of knowing which medication one is receiving. Since both drugs probably are perceived as positive treatment options in MS today it is unlikely that there will be a predominant placebo effect of either of the treatment options.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Relapsing Remitting MS according to the 2017 revised McDonald cri-teria 27 OR one demyelinating episode in conjunction with at least one asympto-matic high intensity T2 lesion with size and location compatible with MS.
* Untreated OR treated with first-line injectables (interferon or glatiramer acetate)
* Between the age of 18 and 50 years (inclusive) of age
* No more than ten years of disease duration
* During the previous year, clinical or radiological disease activity defined as at least one of the following:

  * ≥ 1 relapse
  * ≥ 2 T2 lesions
  * ≥ 1 Gd+ lesions
* Expanded Disability Status Scale: 0 - 5,5 (inclusive)
* In fertile females, willing to comply with effective contraceptive methods. These include birth control pills, surgical sterilization of patient or partner or intrauterine device. Non-fertile women is defined as more than 12 months of amenorrhea without an alternative medical cause or, in case of ambiguities, an follicle stimulation hormone level in the postmenopausal range.

Exclusion Criteria:

* Diagnosis of Progressive MS
* Pregnant or lactating women: human chorionic gonadotropin (s-HCG) will be tested on all women at screening, before each study-related infusion and in any situation where there is a reason to suspect pregnancy during the trial, eg delayed menstrual period more than five days above expected time.
* Patients having contraindication for or otherwise not compliant with MRI investigations
* Simultaneous treatment with other immunosuppressive drugs
* Active, severe infections Signs of infections are assessed before inclusion and each study-related infusion through clinical examination and further evaluated by laboratory and other relevant investigations in case of suspected ongoing infection. Hepatitis serology (HBsAg and anti-HBc) will be evaluated before treatment onset.
* Severe cardiac disorder, eg signs of congestive heart failure or coronary artery disease. This will be evaluated through clinical assessment before inclusion.
* Vaccination within 4 weeks of first dose of study medication.
* Documented allergy or intolerance to any of the investigational products.
* Severe psychiatric condition

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2021-07 (Actual); Study Completion 2021-08 (Actual)

PRIMARY OUTCOMES:
Freedom of relapse | Within 2 years
  The relative risk of experiencing a relapse during the two-year period for either compound.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Svenningsson, MD, PhD, Principal Investigator — Dept.of Medicine, Sect.of Neurology, Danderyd Hospital
Locations (17):
- Sweden (17):
  - South Älvsborg Hospital, Borås
  - Falun Hospital, Falun
  - Gävle Hospital, Gävle
  - Saghlgrenska Hospital, Gothenburg
  - Helsingborg Hospital, Helsingborg
  - Karlstad Hospital, Karlstad
  - Halland Hospital Kungsbacka, Kungsbacka
  - Linköping University Hospital, Linköping
  - Nyköping Hospital, Nyköping
  - Örebro University Hospital, Örebro
  - Östersund Hospital, Östersund
  - Capio StGöran Hospital, Stockholm
  - Danderyd hospital, Stockholm
  - Fredrik Piehl, Stockholm
  - Karolinska Hospital Huddinge, Stockholm
  - Umeå University, Umeå
  - Uppsala Academiska Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Svenningsson A, Frisell T, Burman J, Salzer J, Fink K, Hallberg S, Hambraeus J, Axelsson M, Nimer FA, Sundstrom P, Gunnarsson M, Johansson R, Mellergard J, Rosenstein I, Ayad A, Sjoblom I, Risedal A, de Flon P, Gilland E, Lindeberg J, Shawket F, Piehl F, Lycke J. Safety and efficacy of rituximab versus dimethyl fumarate in patients with relapsing-remitting multiple sclerosis or clinically isolated syndrome in Sweden: a rater-blinded, phase 3, randomised controlled trial. Lancet Neurol. 2022 Aug;21(8):693-703. doi: 10.1016/S1474-4422(22)00209-5. PMID 35841908